CLINICAL TRIAL: NCT05098964
Title: Physical Activity in COPD
Brief Title: Pedometer Assisted Physical Activity in Individuals With COPD. A Multicenter Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yusup subagio sutanto (Other)
Responsible Party: Sponsor-Investigator, Yusup subagio sutanto, Chief of pulmonary department, Universitas Sebelas Maret
Organization: Universitas Sebelas Maret (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 713/IX/HREC/2018
Record Dates: First submitted 2021-10-17; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pulmonary rehabilitation; Tele-medicine; Exercise capacity; Dyspnoea; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (pedometer) (Experimental): Participants received an Omron HJ 321 pedometer (Omron Healthcare Co Ltd, Kyoto, Japan) and were asked to walk at home at the fastest step pace as possible, for at least 30 minutes every day, up to 6 weeks.
  Interventions: Device: pedometer home based rehabilitation
- Control Group (Experimental): participants received supervised exercise training at outpatient clinics for total 18 sessions (3 weekly sessions for 6 weeks).
  Interventions: Other: Exercise training

INTERVENTIONS:
Device: pedometer home based rehabilitation — Home based pulmonary rehabilitation for 6 weeks using pedometer Omron HJ 321 pedometer (Omron Healthcare Co Ltd, Kyoto, Japan)
  Other Names: pedometer
  Arms: Study Group (pedometer)
Other: Exercise training — Hospital based exercise training for 6 weeks
  Arms: Control Group

SUMMARY:
Home based and tele-rehabilitation programs may be potentially useful to deliver and to maintain the benefits in difficult-to-reach areas. Tele-health technologies allow for distribution of healthcare services and exchange of information between healthcare providers and patients in different geographical locations and provide an important tool to reach people living in rural communities. In a previous single center study, we had shown that a home pedometer assisted program to enhance physical activity was as effective as and cheaper than a standard outpatient supervised exercise training program.13 We wondered whether the results of that study 13 might be confirmed in a larger multicenter randomized controlled trial (RCT). Therefore the aim of this multicenter RCT was to evaluate the benefits and costs of a program of pedometer assisted physical activity as compared to standard hospital outpatient supervised exercise training program.

DETAILED DESCRIPTION:
A multicenter RCT was conducted in Moewardi (Surakarta, Central Jawa, Indonesia) and Mohammad Rabain (Muara Enim, South Sumatra, Indonesia) hospitals from February the 1st, 2019 to February the 29th 2020. The study was performed according to the Helsinki Declaration, approved by the Committee of Moewardi Hospital, Surakarta, Central Jawa, Indonesia (Number 713/IX/HREC/2018, September 26th, 2018 and Indonesian Ministry of Health).Participants with COPD as defined by the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guidelines and eligible for this study were allocated into two groups using a randomly generated sequence. Before and after the program, the following outcome measures; 6MWT, BODE, physical activity, MRC and CAT Score.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with COPD as defined by the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guidelines,2 40-80 years old, were recruited from the outpatient clinics of Moewardi and Mohammad Rabain hospitals.
* All subjects had to be in stable conditions as assessed by absence of worsening in symptoms, i.e. no change in cough, and/or sputum beyond day-to-day variability which would have been sufficient to warrant a change in the management prescribed at discharge from hospitals or prescribed at home by their GP, and stability in blood gas values (e.g. no respiratory acidosis).

Exclusion Criteria:

* Individuals refusing to participate, participated in a pulmonary rehabilitation program during the previous 6 months, or with active malignancy, previous lung surgery, unstable cardiovascular diseases, orthopaedic and/or neuromuscular diseases interfering with their ability to walk, or inability to connect with internet and operate WhatsApp video call applications were excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Exercise Tolerance | Before and after program (6 weeks)
  Exercise tolerance was assessed by mean of the 6MWT according to accepted

SECONDARY OUTCOMES:
Physical Activity | Before and after program (6 weeks)
  Physical activity was measured as daily steps, based on an average step count of 7 days obtained from the pedometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary department of medical faculty Universitas Sebelas Maret, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided